## **Study Title:** A Prospective Randomized Study on the Immediate Loading of Mandibular Overdentures Supported by a Parallel Sided or Tapered Dental Titanium Implant

NCT#: 03272828

Principal Investigator: Mats Kronstrom, DDS, PhD

Document Name: Statistical Analysis Plan

Approval Date: 12/14/2023

## **Statistical Analysis Plan**

The proportions of implant failures in the two treatment groups were reported. A test of the hypotheses of no difference between failure proportions was conducted using Fisher's exact test. For the ISQ and bone loss outcomes, means and standard deviations were reported at each visit. Unequal-variance 2-sample t-tests were used to compare group means for the 60-month outcomes.